CLINICAL TRIAL: NCT03240874
Title: SweetMama Usability and Feasibility: Testing of a Novel Technology for Diabetes Education and Support to Pregnant Women
Brief Title: SweetMama: Testing of a Novel Technology for Diabetes Education and Support to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00205409; 1R21HD094271-01 (NIH); 5R21HD094271-02 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes; Diabetes Type 2 in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Two phases of study:
  1. Usability testing - focus groups followed by individual usability testing (single arm)
  2. Feasibility testing - pilot randomized controlled trial of SweetMama care versus usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usability - Focus Group (Experimental): Mobile Application Usability Testing: SweetMama Focus Groups
  Focus groups: Women with a confirmed intrauterine pregnancy or postpartum until 12 weeks after delivery with gestational diabetes mellitus or type 2 diabetes mellitus will be recruited to undergo a single 1-hour focus group.
  Interventions: Behavioral: SweetMama Focus Groups
- Usability - Individual Testing (Experimental): Mobile Application Usability Testing: SweetMama Individual Testing
  Individual testing: Women with a confirmed intrauterine pregnancy (any gestational age) or who are up to 4 weeks postpartum, with gestational diabetes mellitus or type 2 diabetes mellitus, will be recruited to use SweetMama for 2 weeks and provide feedback.
  Interventions: Behavioral: SweetMama Individual Testing
- Feasibility - Pilot Randomized Trial, SweetMama arm (Experimental): Mobile Application Feasibility Testing: SweetMama Pilot Trial, SweetMama arm
  Women recruited to the pilot RCT phase will enroll in the study upon initiation of prenatal care for diabetes, which could be early in pregnancy at the time of first prenatal visit, or at a later point if they have transferred care to this site. Women randomized to receive SweetMama care will be oriented to use of SweetMama and will then use the intervention (messages, library, goal setting, and appointment reminders) throughout pregnancy and the first 8 weeks postpartum, at which point they will undergo surveys and interviews.
  Interventions: Behavioral: SweetMama Feasibility Testing - Pilot Randomized Trial
- Feasibility - Pilot Randomized Trial, usual care arm (No Intervention): Mobile Application Feasibility Testing: SweetMama Pilot Trial, usual care arm
  Women recruited to the pilot RCT phase will enroll in the study upon initiation of prenatal care for diabetes, which could be early in pregnancy at the time of first prenatal visit, or at a later point if they have transferred care to this site. Women randomized to usual care will be undergo entry and exit surveys (at 6-8 weeks postpartum) but will not interact with SweetMama.

INTERVENTIONS:
Behavioral: SweetMama Focus Groups — Focus groups will assess tool functionality, design, interpretability, and acceptability (initial reaction, attitude, and receptiveness) of SweetMama via qualitative interviewing. The group format will generate feedback on areas that may not be revealed in a one-on-one interview.
  Arms: Usability - Focus Group
Behavioral: SweetMama Individual Testing — Women will be oriented to SweetMama use on their own Android- or Apple-based phones. The goals of this phase are to collect data from diverse users that will (1) confirm that the mobile apps are functioning (not crashing) across a wide range of devices and operating systems, (2) provide basic information about app usage and user satisfaction (3) inform the development of future iterations by analyzing participant characteristics and use, and (4) collect quality assurance data that will allow the research team to refine the applications. Women will use SweetMama for 2 weeks, engage in periodic "check-ins" with the research assistant, and participate in a semi-structured interview upon completion of SweetMama usage.
  Arms: Usability - Individual Testing
Behavioral: SweetMama Feasibility Testing - Pilot Randomized Trial — Women will be oriented to SweetMama use on their own Android- or Apple-based phones. The goals of this phase are to collect data from diverse users that will determine acceptability, feasibility, and pilot procedures in anticipation of a fully powered randomized controlled trial. Women will use SweetMama from enrollment (early pregnancy) to up to 8 weeks postpartum, engage in periodic "check-ins" with the research assistant, and participate in surveys and a semi-structured interview upon completion of SweetMama usage.
  Arms: Feasibility - Pilot Randomized Trial, SweetMama arm

SUMMARY:
Diabetes during pregnancy is a challenging clinical situation requiring substantial patient engagement. The investigators have developed a novel early-phase tool, called SweetMama, that incorporates educational, motivational and supportive elements to positively impact maternal health behaviors. This phase of work involves develop an optimized version of SweetMama via a 2-step sequential process of in-depth usability and feasibility testing. First the investigators will conduct focus groups and individual usability testing followed by refinement of SweetMama based on participant input. Next, the investigators will conduct feasibility testing via a pilot randomized trial to determine acceptability, feasibility, and pilot procedures for a fully powered larger trial.

DETAILED DESCRIPTION:
In prior work, the investigators created a text messaging curriculum that was well-received by patients for diabetes-related education and support during pregnancy. The team has now drawn upon these earlier phases to develop a mobile health behavior tool to educate and support low-income, minority pregnant women with Gestational Diabetes Mellitus and Type 2 Diabetes Mellitus. This "first-of-its-kind" mHealth platform for pregnant women with GDM or T2DM is called SweetMama. SweetMama is a theory-driven application that delivers an interactive, goal-oriented educational and motivational diabetes-focused curriculum. SweetMama currently functions as a user-friendly application in which participants are delivered curriculum messages and have the opportunity to receive novel educational, motivational, or supportive content when desired by patients; they additionally have the opportunity to view library content and receive support with goal-setting.

To perform usability testing, the investigators will first conduct focus groups with 10-20 low-income pregnant women with diabetes to evaluate tool functionality, design, and interpretability. The investigators will then conduct a phase of individual usability testing with 20 women, who will use SweetMama for 2 weeks followed by qualitative (interviews) and quantitative (questionnaires and user interaction data) assessments of tool satisfaction and use.

Next, to perform feasibility testing, the investigators will recruit approximately 40 low-income pregnant women with diabetes to be randomized to either usual care or SweetMama care, from the beginning of their enrollment at this clinical site for diabetes-specific prenatal care through the first 8 weeks postpartum. Randomization will be unbalanced to favor receipt of the intervention. Participants will undergo surveys and interviews at multiple time points, and those who are randomized to experience SweetMama will undergo an exit interview. Outcomes will include retention, treatment adherence, functionality of the tool, and user interactivity with the tool. The expected outcome of the pilot RCT phase is a better understanding of feasibility of a SweetMama trial via field testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Gestational diabetes mellitus or type 2 diabetes mellitus
* English-speaking
* Gestational age
* Focus groups: Confirmed intrauterine pregnancy at least 8 weeks' gestational age or postpartum until 12 weeks after delivery
* Individual testing: Confirmed intrauterine pregnancy prior to 30 weeks' gestational age
* Pilot trial: Confirmed intrauterine pregnancy prior to 30 weeks' gestational age
* Low income, defined as use of publicly-supported insurance for prenatal care or household income <200% of poverty line for family size
* Access to a mobile smartphone ( for longitudinal testing phase)

Exclusion Criteria:

* Failure to meet the inclusion criteria above
* Non-viable pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Yee, MD, MPH, Principal Investigator — Assistant Professor, Maternal and Fetal Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez H, DiTosto JD, Niznik CM, Yee LM. Understanding Food Security as a Social Determinant of Diabetes-Related Health during Pregnancy. Am J Perinatol. 2023 Jun;40(8):825-832. doi: 10.1055/s-0041-1740194. Epub 2021 Nov 28. PMID 34839467
- [Result] Leziak K, Birch E, Jackson J, Strohbach A, Niznik C, Yee LM. Identifying Mobile Health Technology Experiences and Preferences of Low-Income Pregnant Women with Diabetes. J Diabetes Sci Technol. 2021 Sep;15(5):1018-1026. doi: 10.1177/1932296821993175. Epub 2021 Feb 19. PMID 33605158
- [Result] Jackson J, Leziak K, Niznik CM, Yee LM. Health Care Providers' Utilization of and Perspectives on Mobile Health Technology for Diabetes and Pregnancy Support. Diabetes Spectr. 2021 Aug;34(3):257-267. doi: 10.2337/ds20-0040. Epub 2021 Mar 9. PMID 34511852
- [Result] Yee LM, Leziak K, Jackson J, Strohbach A, Saber R, Niznik CM, Simon MA. Patient and Provider Perspectives on a Novel Mobile Health Intervention for Low-Income Pregnant Women With Gestational or Type 2 Diabetes Mellitus. J Diabetes Sci Technol. 2021 Sep;15(5):1121-1133. doi: 10.1177/1932296820937347. Epub 2020 Jul 5. PMID 32627582
- [Result] Steinberg JR, Yeh C, Jackson J, Saber R, Niznik CM, Leziak K, Yee LM. Optimizing Engagement in an mHealth Intervention for Diabetes Support During Pregnancy: the Role of Baseline Patient Health and Behavioral Characteristics. J Diabetes Sci Technol. 2022 Nov;16(6):1466-1472. doi: 10.1177/19322968211035441. Epub 2021 Aug 22. PMID 34423677
- [Result] Yee LM, Leziak K, Jackson J, Niznik CM, Simon MA. Health Care Providers' Perspectives on Barriers and Facilitators to Care for Low-Income Pregnant Women With Diabetes. Diabetes Spectr. 2020 May;33(2):190-200. doi: 10.2337/ds19-0044. PMID 32425457
- [Result] Birch EM, Leziak K, Jackson J, Dahl E, Niznik CM, Yee LM. Content Quality of YouTube Videos About Gestational Diabetes: Systematic Evaluation. JMIR Diabetes. 2022 Apr 7;7(2):e30156. doi: 10.2196/30156. PMID 35389355
- [Derived] Roytman MV, Lu L, Soyemi E, Leziak K, Niznik CM, Yee LM. Exploring Psychosocial Burdens of Diabetes in Pregnancy and the Feasibility of Technology-Based Support: Qualitative Study. JMIR Diabetes. 2025 Apr 21;10:e53854. doi: 10.2196/53854. PMID 40258264

RESULTS

PARTICIPANT FLOW:
Groups:
- Usability - Focus Group: Mobile Application Usability Testing: SweetMama Focus Groups
  Focus groups: Women with a confirmed intrauterine pregnancy or postpartum until 12 weeks after delivery with gestational diabetes mellitus or type 2 diabetes mellitus will be recruited to undergo a single 1-hour focus group.
  SweetMama Focus Groups: Focus groups will assess tool functionality, design, interpretability, and acceptability (initial reaction, attitude, and receptiveness) of SweetMama via qualitative interviewing. The group format will generate feedback on areas that may not be revealed in a one-on-one interview.
- Usability - Individual Testing: Mobile Application Usability Testing: SweetMama Individual Testing
  Individual testing: Women with a confirmed intrauterine pregnancy (any gestational age) or who are up to 4 weeks postpartum, with gestational diabetes mellitus or type 2 diabetes mellitus, will be recruited to use SweetMama for 2 weeks and provide feedback.
  SweetMama Individual Testing: Women will be oriented to SweetMama use on their own Android- or Apple-based phones. The goals of this phase are to collect data from diverse users that will (1) confirm that the mobile apps are functioning (not crashing) across a wide range of devices and operating systems, (2) provide basic information about app usage and user satisfaction (3) inform the development of future iterations by analyzing participant characteristics and use, and (4) collect quality assurance data that will allow the research team to refine the applications. Women will use SweetMama for 2 weeks, engage in periodic "check-ins" with the research assistant, and participate in a semi-structured interview upon completion of SweetMama usage.
- Feasibility - Pilot Randomized Trial, SweetMama Arm: Mobile Application Feasibility Testing: SweetMama Pilot Trial, SweetMama arm
  Women recruited to the pilot RCT phase will enroll in the study upon initiation of prenatal care for diabetes, which could be early in pregnancy at the time of first prenatal visit, or at a later point if they have transferred care to this site. Women randomized to receive SweetMama care will be oriented to use of SweetMama and will then use the intervention (messages, library, goal setting, and appointment reminders) throughout pregnancy and the first 8 weeks postpartum, at which point they will undergo surveys and interviews.
  SweetMama Feasibility Testing - Pilot Randomized Trial: Women will be oriented to SweetMama use on their own Android- or Apple-based phones. The goals of this phase are to collect data from diverse users that will determine acceptability, feasibility, and pilot procedures in anticipation of a fully powered randomized controlled trial. Women will use SweetMama from enrollment (early pregnancy) to up to 8 weeks postpartum, engage in periodic "check-ins" with the research assistant, and participate in surveys and a semi-structured interview upon completion of SweetMama usage.
Period: Overall Study
Arm/Group | Usability - Focus Group | Usability - Individual Testing | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Started | 16 | 24 | 30 | 10
Completed | 16 | 22 | 26 | 9
Not Completed | 0 | 2 | 4 | 1
Not completed — Lost to Follow-up | 0 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usability - Focus Group | Usability - Individual Testing | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm | Total
Number analyzed (Participants) | 16 | 24 | 30 | 10 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] — The usability and feasibility phases did not occur at the same time so age was not analyzed together.
  Years | 33 (6) | 32.07 (5.32) | 31.35 (4.73) | 31.30 (6.91) | 31.89 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 30 | 10 | 80
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 12 | 2 | 25
  Not Hispanic or Latino | 14 | 15 | 18 | 8 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 11 | 20 | 8 | 53
  White | 0 | 4 | 2 | 0 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 9 | 7 | 2 | 20
Region of Enrollment [Number; unit: participants]
  United States | 16 | 24 | 30 | 10 | 80
Diabetes diagnosis [Count of Participants; unit: Participants]
  Gestational diabetes | 8 | 12 | 18 | 7 | 45
  Type 2 diabetes | 8 | 12 | 12 | 3 | 35
Publicly funded insurance [Count of Participants; unit: Participants]
  Yes | 16 | 15 | 25 | 8 | 64
  No | 0 | 9 | 5 | 2 | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — For the usability phase qualitative (interviews) and quantitative (questionnaires and user interaction data) were collected. The focus group, individual usability testing, and feasibility pilot phase were analyzed separately. BMI was collected for the individual usability phase and the feasibility phase. BMI was not collected for the usability focus group. No demographics were collected to determine BMI. Population: BMI was collected for the individual usability phase and the feasibility phase. For the usability focus group, no participants were analyzed for BMI and no data was collected.
  kg/m^2
    number analyzed (Participants) | 0 | 24 | 30 | 10 | 64
    (all) |  | 37.20 (8.08) | 42.94 (12.40) | 36.67 (9.03) | 39.81 (10.86)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Identifying Themes on SweetMama Features
Description: Participants completed qualitative group interviews to yield information about SweetMama features and participant preferences after use in the usability laboratory. The identified themes are outlined, and the criteria used to determine the outcome measure is the number of participants who endorsed each theme related to SweetMama features.
Time Frame: 60-90 minutes
Population: Focus group participants with confirmed diagnosis of Gestational Diabetes or Type 2 Diabetes. We recorded the identified themes and the number of participants who expressed each theme.
Measure: Count of Participants; unit: Participants
Arm/Group | Usability - Individual Testing
Number analyzed (Participants) | 16
Participants
  Visual features personalized | 9
  Aesthetic appeal | 11
  Content organization | 11
  Content is practical and helpful | 2
  Goal-setting activity | 4
  Option to "favorite" | 3
  Interactivity of messages | 1

2. Primary Outcome: Number of Participants Who Used the SweetMama Application
Description: Feasibility will be assessed as both ability to recruit and retain participants and as a percentage of active SweetMama use. Feasibility targets for study retention will be set at 80% retention; the feasibility target for SweetMama adoption will be 80% active use (at least weekly interaction with SweetMama content).
Time Frame: After 8 weeks postpartum (approximately 18-38 weeks of enrollment)
Population: Participants assigned to use the SweetMama application or usual care.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 30 | 10
Participants
  Retention | 26 | 9
  Ever used application | 30 | 0
  Used application at least once/week during pregnancy | 30 | 0
  Used application at least once/week during postpartum | 26 | 0

3. Secondary Outcome: Usage Time of SweetMama Application
Description: User interaction with the SweetMama application for the total usage time of the application in minutes was assessed at two timepoints. In the individual usability phase, total usage time of the application was evaluated after 2 weeks of enrollment. In the feasibility phase, total usage time of the application was evaluated after 8 weeks postpartum. The reported number is minutes of use which is a total number of minutes of usage time after 2 weeks of enrollment and after 8 weeks postpartum.
Time Frame: After 2 weeks of enrollment (individual usability phase) and after 8 weeks postpartum (feasibility trial; approximately 18-38 weeks of enrollment)
Population: Participants enrolled to engage with the SweetMama application in both Aim 1 and Aim 2. For usability testing, N= 23 because one participant never opened the application which removes the participant from the analysis population of this outcome.
Measure: Median (Inter-Quartile Range); unit: minutes of SweetMama use
Arm/Group | Usability - Individual Testing | Feasibility - Pilot Randomized Trial, SweetMama Arm
Number analyzed (Participants) | 23 | 30
minutes of SweetMama use | 20.5 [11.53 to 27.93] | 48.53 [23.53 to 69.90]

4. Secondary Outcome: Usability Testing of SweetMama Application With the System Usability Scale Survey
Description: Usability of SweetMama will be assessed using the System Usability Scale min 0 max 100
  1=Acceptable(>70) 2=Marginal(50<SUS<=70) 3=Not Acceptable(<=50) Usability testing of the SweetMama application with System Usability Scale was assessed at two timepoints. In the individual usability phase, usability testing was evaluated after 2 weeks of enrollment. In the feasibility phase, usability testing was evaluated after 8 weeks postpartum.
Time Frame: as for outcome 3
Population: In the individual usability phase, 22 participants completed the USE Questionnaire; 2 missing for non-user of application and loss to follow-up.
  In the feasibility phase, 28 participants completed the USE Questionnaire; 2 missing for loss to follow-up and did not deliver at site hospital.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usability - Individual Testing | Feasibility - Pilot Randomized Trial, SweetMama Arm
Number analyzed (Participants) | 22 | 28
score on a scale | 75.00 [60.00 to 87.50] | 85.00 [70.00 to 88.75]

5. Secondary Outcome: Usability Testing of SweetMama Application With the Useful, Satisfaction and Ease of Use Questionnaire
Description: Usability of SweetMama will be assessed using the Usefulness, Satisfaction and Ease of Use (USE) Questionnaire. The higher the participant scored means the participant did better.
  Usefulness: (sum(use_1 - use_8)/56)*100, range from 14.29 to 100 Satisfaction: (sum(use_24-use_30)/49)*100, range from 14.29 to 100 Ease of Use (USE): (sum(use_9-use_19)/77)*100, range from 14.29 to 100 Usability testing of the SweetMama application was assessed at two timepoints. In the individual usability phase, usability testing was evaluated after 2 weeks of enrollment. In the feasibility phase, usability testing was evaluated after 8 weeks postpartum.
Time Frame: After 2 weeks of enrollment (individual usability phase) and after 8 weeks postpartum (feasibility trial; approximately 18-38 weeks of enrollment))
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usability - Individual Testing | Feasibility - Pilot Randomized Trial, SweetMama Arm
Number analyzed (Participants) | 22 | 28
score on a scale
  Usefulness | 83.93 [64.29 to 94.64] | 82.14 [71.43 to 85.71]
  Ease of use | 85.71 [83.12 to 97.40] | 88.31 [84.42 to 94.81]
  Ease of Learning | 87.50 [85.71 to 100.00] | 91.07 [85.71 to 100.00]
  Satisfaction | 85.71 [69.39 to 100.00] | 82.65 [73.47 to 93.88]

6. Secondary Outcome: Diabetes Self-efficacy
Description: Diabetes self-efficacy measured via patient-reported outcomes (Diabetes Empowerment Scale), which is scored from 8 to 40 (sum of individual items), where higher total scores indicate higher self-efficacy
Time Frame: After 8 weeks postpartum (approximately 18-38 weeks of enrollment)
Population: In SweetMama arm, 28 completed the Diabetes self-efficacy measure at delivery; 2 missing for loss to follow-up and not delivered at site hospital.
  In the SweetMama arm, 27 completed Diabetes self-efficacy measure postpartum; 3 missing for not delivered at site hospital and 2 lost to follow-up.
  In the usual care arm, 9 completed Diabetes self-efficacy measure postpartum; 1 missing for pregnancy termination.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 28 | 10
score on a scale
  Diabetes self-efficacy Delivery | 4.44 [4.13 to 4.88] | 3.88 [3.75 to 4.63]
  Diabetes self-efficacy Postpartum: number analyzed (Participants) | 27 | 9
  Diabetes self-efficacy Postpartum | 4.50 [4.13 to 4.88] | 4.50 [4.13 to 4.75]

7. Secondary Outcome: Patient Activation
Description: Patient activation measured patient engagement in healthcare via patient-reported outcomes (Patient Activation Measure), which is scored from 0 to 100 (sum of all scores, scaled to a 0-100-point system), where higher scores indicate greater activation.
Time Frame: After 8 weeks postpartum (approximately 18-38 weeks of enrollment)
Population: In SweetMama arm, 28 completed Patient Activation Measure at delivery; 2 missing for 1 lost to follow-up and 1 participant not delivered at site hospital.
  In the SweetMama arm, 27 completed Patient Activation Measure postpartum; 3 missing for 1 participant not delivered at site hospital and 2 lost to follow-up.
  In the usual care arm, 9 complete Patient Activation Measure postpartum; 1 missing for pregnancy termination.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 28 | 10
score on a scale
  Patient activation Delivery | 84.95 (11.44) | 88.31 (8.24)
  Patient activation Postpartum: number analyzed (Participants) | 27 | 9
  Patient activation Postpartum | 88.55 (8.76) | 93.85 (4.87)

8. Secondary Outcome: Difference in Hemoglobin A1c From Enrollment to Delivery
Description: Hemoglobin A1c will be assessed as a continuous measure reflecting the difference from enrollment to final. A1c before delivery, we controlled for A1c at enrollment and week difference
Time Frame: After 8 weeks postpartum (approximately 18-38 weeks of enrollment)
Population: For feasibility testing, N value differs because 1 participant was lost to follow-up in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 29 | 9
Participants
  Hemoglobin A1c - No change | 3 | 2
  Hemoglobin A1c - Worsened by >1% (got higher) | 10 | 1
  Hemoglobin A1c - Improved by >1% (lower) | 16 | 6

9. Other Pre Specified Outcome: Clinical Outcomes of Pregnancy - Percentage of Patients With Hypertensive Disorders of Pregnancy
Description: In feasibility testing participants, clinical outcomes include hypertensive disorders of pregnancy.
Time Frame: After delivery (approximately 10-30 weeks of enrollment)
Population: Participants in the feasibility testing- SweetMama application users and usual care participants
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 30 | 10
Participants
  No | 12 | 7
  Yes | 18 | 3

10. Other Pre Specified Outcome: Number of Cesarean Deliveries
Description: In feasibility testing, the mode of delivery was report as number of cesarean deliveries for SweetMama and usual care participants.
Time Frame: After delivery (approximately 10-30 weeks of enrollment)
Population: In the usual care arm, 1 missing for pregnancy termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 30 | 9
Participants | 16 | 4

11. Other Pre Specified Outcome: Clinical Outcomes of Pregnancy - Neonatal Birthweight
Description: In feasibility testing participants, clinical outcomes include neonatal birthweight.
Time Frame: After delivery (approximately 10-30 weeks of enrollment)
Population: SweetMama application participants and usual care participants. N=31 in SweetMama arm due to one set of twins. N=9 in the usual care arm due to pregnancy termination.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 31 | 9
grams | 3089.13 (621.45) | 3042.33 (656.68)

12. Other Pre Specified Outcome: Clinical Outcomes of Pregnancy - Number of Babies With Neonatal Hypoglycemia
Description: In feasibility testing participants, clinical outcomes include neonatal hypoglycemia, (<40 mg/dL).
Time Frame: After delivery (approximately 10-30 weeks of enrollment)
Population: N=9 in the usual care arm due to pregnancy termination.
Measure: Number; unit: number of babies
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 30 | 9
number of babies | 5 | 1

13. Other Pre Specified Outcome: Clinical Outcomes of Pregnancy - Number of Babies With Neonatal Intensive Care Unit Admission
Description: In feasibility testing participants, clinical outcomes include neonatal intensive care unit admission.
Time Frame: After delivery (approximately 10-30 weeks of enrollment)
Population: as for outcome 11
Measure: Number; unit: number of babies
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
Number analyzed (Participants) | 31 | 9
number of babies | 13 | 4

ADVERSE EVENTS:
Time Frame: from participant enrollment to after 8 weeks postpartum (approximately 18-38 weeks of enrollment)
Description: Study specific adverse events definitions were created based on FDA criteria. All events were unrelated to the study. The usability phase and feasibility phases were conducted separately and adverse events were not monitored at all for the usability phase and not included in this section. Adverse events were assessed for only participants related to the prenatal and postpartum periods which include events related to the labor and delivery or the immediate postpartum hospitalization.
Arm/Group | Feasibility - Pilot Randomized Trial, SweetMama Arm | Feasibility - Pilot Randomized Trial, Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 9/30 | 2/10
Other Adverse Events (participants affected / at risk) | 10/30 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feasibility - Pilot Randomized Trial, SweetMama Arm (N=30) | Feasibility - Pilot Randomized Trial, Usual Care Arm (N=10)
Unanticipated hospital admission requiring medical or surgical intervention for life-threatening eve (Infections and infestations) | 1 (1) | 0 (0)
Unanticipated hospital admission requiring medical or surgical intervention for life-threatening eve (Hepatobiliary disorders) | 1 (1) | 0 (0)
Unanticipated hospital admission requiring medical or surgical intervention for life-threatening eve (Renal and urinary disorders) | 1 (1) | 0 (0)
Preterm birth <34 weeks of gestation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Unanticipated hospital admission requiring medical or surgical intervention for life-threatening eve (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Unanticipated hospital admission requiring medical or surgical intervention for life-threatening eve (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Neonatal intensive care unit admission for pressor support, ventilator support, or anti-seizure medi (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Only participants of infants with neonatal intensive care unit admission for pressor support, ventilator support, or anti-seizure medicine are considered as having adverse events. NICU admissions for other reasons were not considered in this section
Maternal intensive care unit admission (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feasibility - Pilot Randomized Trial, SweetMama Arm (N=30) | Feasibility - Pilot Randomized Trial, Usual Care Arm (N=10)
Hospital admission requiring medical intervention or observation for a diabetes-related indication (Endocrine disorders) | 4 (7) | 3 (3)
Preterm birth ≥34 weeks of gestation (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03240874/Prot_SAP_002.pdf
  • Informed Consent Form: Focus Group Usability Testing (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03240874/ICF_003.pdf
  • Informed Consent Form: Individual Usability Testing (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03240874/ICF_004.pdf